CLINICAL TRIAL: NCT04051944
Title: An Open-Label Extension Study to Investigate the Long-Term Safety, Tolerability, and Efficacy of Rozanolixizumab in Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: A Study to Assess Long-term Safety, Tolerability and Efficacy of Rozanolixizumab in Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIDP04; 2018-004392-12 (EudraCT Number)
Expanded Access: NCT05014724 (No longer available)
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Keywords: Chronic inflammatory demyelinating polyradiculoneuropathy; CIDP; UCB7665; rozanolixizumab
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rozanolixizumab (Experimental): Subjects in this arm will receive predefined subcutaneous doses of rozanolixizumab at a specified frequency.
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Subjects will receive rozanolixizumab in a specified sequence during the treatment period.

SUMMARY:
The purpose of the study is to assess long-term safety and tolerability of weekly doses of rozanolixizumab in subjects with chronic inflammatory demyelinating polyradiculoneuropathy (CIDP).

ELIGIBILITY:
Inclusion Criteria:

* Subject who has completed one of the previous rozanolixizumab study(ies) that allow access to the present study (e.g. study CIDP01)
* Female subjects of childbearing potential must agree to use a highly effective method of birth control, during the study and for a period of 3 months after their final dose of investigational medicinal product (IMP)
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active during the study and for 3 months after the final administration of IMP

Exclusion Criteria:

* Subject has any medical (acute or chronic illness) or psychiatric condition that, in the opinion of the investigator, could harm the subject or would compromise the subject's ability to participate in this study
* Subject has a clinically relevant active infection (eg, sepsis, pneumonia, abscess)
* Subject has a known hypersensitivity to any components of rozanolixizumab
* Subject intends to have a live vaccination during the course of the study or within 7 weeks following the final dose of rozanolixizumab
* Subject has an ongoing serious adverse event (SAE) or a medical condition in the parent study that the investigator considers to put the subject at a significantly increased risk of participating in CIDP04
* Subject has any planned elective surgery due to occur during the study dosing period which in the opinion of the investigator could interfere with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (14):
- United States (4):
  - Cidp04 50082, Scottsdale, Arizona
  - Cidp04 50075, Augusta, Georgia
  - Cidp04 50117, Charlotte, North Carolina
  - Cidp04 50080, Durham, North Carolina
- Belgium (3):
  - Cidp04 40169, Ghent
  - Cidp04 40002, Leuven
  - Cidp04 40120, Liège
- Cidp04 40126, Copenhagen, Denmark
- Cidp04 40170, Strasbourg, France
- Germany (2):
  - Cidp04 40134, Essen
  - Cidp04 40140, Göttingen
- Cidp04 40034, Amsterdam, Netherlands
- Cidp04 40160, Barcelona, Spain
- Cidp04 40167, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

REFERENCES:
- [Derived] Querol L, De Seze J, Dysgaard T, Levine T, Rao TH, Rivner M, Hartung HP, Kiessling P, Shimizu S, Marmol D, Bozorg A, Colson AO, Massow U, Eftimov F; CIDP01 Study Investigators. Efficacy, safety and tolerability of rozanolixizumab in patients with chronic inflammatory demyelinating polyradiculoneuropathy: a randomised, subject-blind, investigator-blind, placebo-controlled, phase 2a trial and open-label extension study. J Neurol Neurosurg Psychiatry. 2024 Aug 16;95(9):845-854. doi: 10.1136/jnnp-2023-333112. PMID 38729747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in Aug 2019 and concluded in Nov 2021.
Pre-assignment Details: Participant Flow refers to the Enrolled Set. Participants from parent study CIDP01 (NCT03861481) who had completed the Treatment Period without a relapse of chronic inflammatory demyelinating polyradiculoneuropathy were directly enrolled into this study. Newly treated participants are participants treated with placebo in parent study CIDP01 (NCT03861481). Previously treated participants are participants treated with rozanolixizumab in parent study CIDP01 (NCT03861481).
Groups:
- Rozanolixizumab (Newly Treated); Rozanolixizumab (Previously Treated): Participants received rozanolixizumab Dose A as a subcutaneous infusion once weekly up to Week 76.
Period: Overall Study
Arm/Group | Rozanolixizumab (Newly Treated) | Rozanolixizumab (Previously Treated)
Started | 11 | 10
Completed | 3 | 6
Not Completed | 8 | 4
Not completed — Study ending | 1 | 1
Not completed — Early study termination by participant | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 3 | 0
Not completed — Adverse event, non- fatal | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Safety Set (SS) which consisted of all enrolled study participants who were administered at least one dose of rozanolixizumab in CIDP04.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rozanolixizumab (Newly Treated) | Rozanolixizumab (Previously Treated) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (5.1) | 59.1 (15.9) | 59.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 8 | 9 | 17
  Other/Mixed | 0 | 1 | 1
  Missing | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 9 | 10 | 19
  Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product, which does not necessarily had a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE was defined as any event that was not present prior the first administration of investigational medicinal product (IMP) in CIDP04 study or any unresolved event already present before the first administration of IMP in CIDP04 study that worsened in intensity following exposure to treatment until 8 weeks following the last administration of IMP in CIDP04 study.
Time Frame: From Baseline until Follow-Up Visit (up to Week 84)
Population: The Safety Set (SS) consisted of all enrolled study participants who were administered at least one dose of rozanolixizumab in CIDP04.
Measure: Count of Participants; unit: Participants
Arm/Group | Rozanolixizumab (Newly Treated) | Rozanolixizumab (Previously Treated)
Number analyzed (Participants) | 11 | 10
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: From Baseline until Follow-Up Visit (up to Week 84)
Description: A TEAE was defined as any event that was not present prior the first administration of IMP in CIDP04 study or any unresolved event already present before the first administration of IMP in CIDP04 study that worsened in intensity following exposure to treatment until 8 weeks following the last administration of IMP in CIDP04 study.
Arm/Group | Rozanolixizumab (Newly Treated) | Rozanolixizumab (Previously Treated)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/10
Other Adverse Events (participants affected / at risk) | 10/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rozanolixizumab (Newly Treated) (N=11) | Rozanolixizumab (Previously Treated) (N=10)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rozanolixizumab (Newly Treated) (N=11) | Rozanolixizumab (Previously Treated) (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (4)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Blood immunoglobulin G decreased (Investigations) | 4 (10) | 4 (8)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (7) | 1 (5)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (2)
Sensory loss (Nervous system disorders) | 2 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04051944/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT04051944/SAP_001.pdf